CLINICAL TRIAL: NCT06515041
Title: Effects of Museum Visits on Neurocognitive Well-being
Acronym: ABC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 24-0031
Record Dates: First submitted 2024-06-26; First posted 2024-07-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MUSEUM VISITS with mediation: group A (Other): This group of volunteers will visit the museum with a mediation (I.E. description of the painting tables by a professional).
  Interventions: Other: brain well-being
- MUSEUM VISITS without mediation: group B (Other): This group of volunteers will visit the museum without a mediation (I.E. description of the painting tables by a professional).
  Interventions: Other: brain well-being
- Control group (Other): This group of volunteers will not visit the museum.
  Interventions: Other: brain well-being

INTERVENTIONS:
Other: brain well-being — Each volunteers will be subjected to an evaluation of his well-being using a previously well established well-being scale, through a list of questions, prior, during and after the visit to the museum. All volunteers will be also equipped with a non invasive NIRS system to measure their emotions (measure of tissus oxygenenation), with a non invasive system of eye tracking glasses to measure where their eyes are looking and with a non invasive system to measure their heart rate.
  Other Names: non invasive Near InfraRed Spectroscopy (NIRS); neon invasive Eye tracking glasses; non invasive Heart rate measurement; Well-being scale (list of questions)

SUMMARY:
The effects of art on health and well-being have been the subject of increasing exploration in recent years. In 2019, the World Health Organization proposed a literature review analyzing the links between art, health (defined as a state of good functioning) and well-being. Currently, the majority of research has focused on populations presenting pathologies (somatic, neurological or psychiatric), very often in older adults. Furthermore, exposure to art (unlike the practice of an artistic activity) still remains under-investigated. However, recent publications (review and longitudinal study) suggest that attending museums would be associated with an increase in well-being, in people with or without pathology.

Supported by the Blood & Brain @ Caen Normandy Scientific Interest Group and the Museum of Fine Arts as part of the Millennium festivities of the city of Caen, the partnership between three Caen laboratories and a Parisian laboratory enabled the drawing of this innovative research which will aim to measure the effects of visiting a museum dedicated to painting on well-being in healthy adults. It will also involve identifying the cerebral, cognitive and socio-emotional processes associated with these effects, via comprehensive and ecologically adapted measurements.

Through understanding the mechanisms specific to exposure to art which promote well-being, this research could have implications for:

1. Promote synergy between cultural and health policies.
2. Design museum experiences as close as possible to human functioning.
3. Open up to new perspectives such as the role of exposure to art in maintaining good health, with the possibility in the longer term of considering research on other arts, other populations, in a lifespan approach.
4. Open up to other studies of the same type involving pairs of patients and caregivers, young people and seniors, etc.

DETAILED DESCRIPTION:
1. Call for volunteers:

   An A5 information poster will be distributed in various structures in the Caen region but also through the press. Participants will be able to contact a member of the research team by email. They will then be contacted in response to this email in order to arrange a telephone appointment. The purpose of this preliminary telephone interview will be to ensure the inclusion criteria without collecting the personal data relating to them. This is to avoid unnecessary travel. If the participant can be included, then a physical appointment will be offered to them in order to carry out the inclusion visit.
2. Inclusion visit:

   An inclusion visit will be carried out during which the participant will be informed of the progress of the study, its implications and their right of withdrawal. A test of the different devices (Near InfraRed Spectroscopy (NIRS), eye-tracking glasses, skin conductance bracelet) under the same conditions as those of the study will be carried out. Then, the participant's consent will be collected via a written form. Finally, the participant will fill out an admission questionnaire with socio-demographic questions, questions related to the aforementioned inclusion criteria, and questions about their cultural practices. Only for participants over 55 years old, an assessment via the Montreal Cognitive Assessment (MoCA - screening tool for mild neurocognitive impairment) will be carried out. At the end of all these acts, the participant will be assigned an inclusion number. The personal data collected will be stored on a single computer at Cyceron.
3. Visit 1 to the Museum of Fine Arts in Caen:

   Experimental groups Participants in the experimental groups will be randomized into two groups: with or without mediation.

   Regardless of their group, they will see the same number of tables. The measurements and questionnaires they will answer will be identical. Upon arrival, participants will be welcomed and then:
   * ● Guided to a room where they will answer well-being and stress questionnaires, and complete cognitive tasks (executive functions, global/local visual attention, episodic memory, empathy and creativity questionnaire).
   * ● Equipped with eye-tracking glasses, the NIRS headband and the bracelet to measure heart rate (electrodermal biosensor bracelets).
   * ● Guided to view 6 paintings. For group A without mediation, participants will be brought in front of each painting and will look at it independently for 2 minutes. For group B with mediation, the mediator, equipped with a lapel microphone, will guide them and explain each painting in 2 minutes. The viewing time and distance will be the same for both groups. After each painting, regardless of the group, participants will indicate the emotions felt by responding on an affect grid.
   * ● Removal of glasses, headband and bracelet.
   * ● After the visit, participants will again answer the questionnaires and the different cognitive tasks, except for the empathy and creativity questionnaires.

   Control group The participants in the control group will visit the museum according to a pre-established route with the same number of paintings as the experimental groups. The duration of viewing each painting will be controlled to be identical to that of the experimental groups, i.e. 2 minutes. On the other hand, they will not wear any device (NIRS, eye tracking and electrodermal bracelet) and will not have mediation. They will answer the same questionnaires and cognitive tasks as the experimental groups: before and after the visit, as well as the affect grid during the visit.
4. Visit 2 to the Museum of Fine Arts in Caen:

For the experimental groups, the changes between visits 1 and 2 will be as follows:

Number of patients

* ● Participants will complete the visit in pairs (composed of 1 member from group A and 1 from group B). These pairs will be divided into two new groups A' (with mediation) and B' (without mediation).
* ● Participants will see 8 paintings (6 paintings already seen during the first + 2 new paintings).

The questionnaires (except empathy and creativity measured only during visit 1), the cognitive tasks and the measurements (oculometric via eye-tracking/ brain activity via NIRS/ cardiac activity (heart rate via the bracelet) will be carried out in the same way as during visit 1.

For the control group:

* ● The procedure for visit 2 will be identical to that of visit 1. As for the experimental groups, only the empathy and creativity questionnaires will not be included in the questionnaires to be completed.
* ● Like the experimental groups, the control group will carry out the visit in pairs (formed from the members of control group C from visit 1).

ELIGIBILITY:
Inclusion Criteria:

* Adults with good mental and brain health
* Participants (18-65 years old inclusive)
* Good brain health: Having a MoCA score (screening tool for mild neurocognitive impairments) of 26 or above for those over 55 years old.
* Fluent in French (native language)
* Person who has given informed consent to participate in the study
* Declare being able to comfortably view a painting during a museum visit without wearing glasses
* Declare being able to listen to a conversation

Exclusion Criteria:

* History or presence of a psychiatric disorder such as mood disorders, psychotic disorders, personality disorders, addictions, that have required or currently require medical follow-up and/or are in an acute phase.
* Mobility difficulties, postural or balance disorders preventing the participant from easily moving around the museum and using stairs
* History or presence of brain injuries such as TBI, stroke, neurological diseases
* Chronic or long-term illnesses that could make standing uncomfortable for the participant
* Taking medication that affects cognitive functioning
* General anesthesia in the past six months
* Vision impairment requiring glasses or resulting in poor detail perception at a distance of 2 to 6 meters
* Person who has visited the permanent collection of the Caen Museum of Fine Arts at least once in the past ten years (Participants are thus either first-time visitors or people who visited the permanent collection more than ten years ago)
* Unable to reach the museum independently
* Hearing impairment (decibel level above 20) not using a hearing aid or whose hearing aid does not sufficiently correct the impairment
* Speech disorder with difficulty communicating with others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of museum visit on wellbeing | before and after the first visit and the second one
  We will use a well established UCL museum wellbeing measures used to assess levels of psychological wellbeing arising from a situation.
Effect of museum visit on eyes tracking | during each visit, 1 and 2
  eyes tracking glasses will be used to evaluate where the volunteers is looking on pictorials
Effect of museum visit on NIRS | during each visit, 1 and 2
  NIRS, non invasive evaluation of frontal brain oxygenation allowing a follow-up of brain emotions
Effet of museum visit on heart rate | during each visit, 1 and 2
  Non invasive evaluation of heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Denis Vivien, phD, Principal Investigator — Caen Normandie University Hospital
Locations (1):
- Caen University Hospital, Caen, France